CLINICAL TRIAL: NCT02862639
Title: Efficacy of Viscosupplementation Associated With Intra-articular Corticosteroid Injection Versus Intra-articular Injection of Corticosteroids Alone in Osteoarthritis of Hip
Acronym: VISCOSUPP-HIP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PA12069
Record Dates: First submitted 2016-08-08; First posted 2016-08-11 (Estimated); Last update posted 2017-07-27 (Actual); Status verified 2016-09

CONDITIONS: Hip Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- injection of viscosupplementation and corticosteroid (Experimental): experimental group
  Interventions: Device: Experimental group
- injection of corticosteroid (Active Comparator): control group
  Interventions: Device: control group

INTERVENTIONS:
Device: Experimental group — patient receive intra articular injection (hip joint) of viscosupplementation in combination with corticosteroid
  Arms: injection of viscosupplementation and corticosteroid
Device: control group — patient receive intra articular injection (hip joint) of corticosteroid alone
  Arms: injection of corticosteroid

SUMMARY:
The current management of osteoarthritis is based on non-pharmacological and pharmacological means which include intra-articular injections.

The recommendations on the management of hip osteoarthritis stipulate that intra-articular injections of corticosteroid may be considered in patients with an exacerbation not responding to oral treatments. Several recent studies show the effectiveness of intra-articular corticosteroids compared with anesthetics. The intra-articular injection of viscosupplementation alone has never been validated in this indication since controlled studies did not show efficacy over placebo. At present, viscosupplementation is considered an anti-osteoarthritic symptomatic slow-acting and its interest is not yet established in hip osteoarthritis.

DETAILED DESCRIPTION:
Show the superiority of intra-articular injection of viscosupplementation in combination with corticosteroid compared to intra-articular injection of corticosteroid alone in the treatment of hip osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* patients with hip osteoarthrosis (stage II et III according Kellgren et Lawrence)
* walking alone patients
* patient consenting to participate to the study
* patient enrolled in the national healthcare insurance program
* patient older than 18 years

Exclusion Criteria:

* Patients with hip osteoarthrosis (stage I et IV according Kellgren et Lawrence)
* patients with rapidly destructive hip osteoarthritis
* patients with inflammatory rheumatism
* patients with microcrystalline arthritis
* patients with hip osteonecrosis
* patients who received corticosteroids during the previous three months
* patients who received a intra articular injection of viscosupplementation during the previous six months
* patient with haemostatic disorder
* patient with consumption of painkillers tier 3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2014-02; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
improving pain | 3 months
  decrease of 20 mm on a visual analog pain scale between the evaluation at day 0 and the evaluation at 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Reims, Reims, France